CLINICAL TRIAL: NCT07165041
Title: Efficacy of Serratus Posterior Superior Intercostal Plane Block in Cardiac Implantable Electronic Device Implantation: A Prospective, Double-Blind, Randomized Controlled Clinical Trial
Brief Title: Efficacy of Serratus Posterior Superior Intercostal Plane Block in Cardiac Device Implantation
Acronym: SPSIPB-CIED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gozde Altun (Other)
Responsible Party: Sponsor-Investigator, Gozde Altun, Lecturer, Department of Anesthesiology and Reanimation, Istanbul University-Cerrahpasa, Cardiology Institute, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1395253
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pain, Postoperative
Keywords: Serratus Posterior Superior Intercostal Plane Block; Cardiac Implantable Electronic Device; Pain Management; Randomized Controlled Trial
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either ultrasound-guided serratus posterior superior intercostal plane (SPSIP) block with local anesthetic or a sham injection with saline. The study is designed as a prospective, double-blind, parallel-group randomized controlled trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers, and outcome assessors will be blinded to group allocation. The block (bupivacaine or sham saline) will be prepared and administered by an anesthesiologist not involved in outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIP Block (Experimental): Ultrasound-guided serratus posterior superior intercostal plane (SPSIP) block performed with 30 mL of 0.25% bupivacaine administered prior to CIED implantation
  Interventions: Procedure: SPSIP Block
- Sham Control (Sham Comparator): Sham procedure with 1 mL saline injection at the same anatomical site, without administration of local anesthetic, prior to CIED implantation.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: SPSIP Block — Ultrasound-guided serratus posterior superior intercostal plane (SPSIP) block performed prior to cardiac implantable electronic device (CIED) implantation. A total of 30 mL of 0.25% bupivacaine will be injected into the interfascial plane between the rhomboid major and serratus posterior superior muscles under sterile conditions.
  Arms: SPSIP Block
Procedure: Sham procedure — Sham procedure with 1 mL saline injection at the same anatomical site, without administration of local anesthetic, prior to CIED implantation.
  Arms: Sham Control

SUMMARY:
This randomized controlled clinical trial investigates the efficacy of the serratus posterior superior intercostal plane block (SPSIPB) in patients undergoing cardiac implantable electronic device (CIED) implantation. Participants will be randomized to receive either SPSIP block with local anesthetic or a sham procedure with saline injection. Pain intensity will be evaluated intraoperatively and at 3, 6, 12, and 24 hours postoperatively using the Visual Analog Scale (VAS). Secondary outcomes include sleep quality at 24 hours assessed with the Sleep Quality Numeric Rating Scale (SQ-NRS), and patient and clinician satisfaction assessed with a 5-point Likert scale. The study is designed as prospective, double-blind, and parallel-group, aiming to improve perioperative pain management in CIED procedures.

DETAILED DESCRIPTION:
Cardiac implantable electronic device (CIED) implantation is a common procedure for the management of arrhythmias and prevention of sudden cardiac death. Although routinely performed under local anesthesia, patients may experience intraoperative and postoperative pain, which can affect hemodynamic stability, recovery, and satisfaction. Effective perioperative analgesia is therefore critical in this patient group, who often present with multiple comorbidities and advanced age. Conventional systemic analgesics may be insufficient or associated with side effects, highlighting the need for alternative approaches.

The serratus posterior superior intercostal plane block (SPSIPB) is a recently described regional anesthesia technique targeting the interfascial plane between the rhomboid major and serratus posterior superior muscles. Previous studies have shown its efficacy in thoracic, breast, clavicular, and minimally invasive cardiac surgeries. However, its role in the context of CIED implantation has not been systematically studied.

This study is designed as a prospective, double-blind, randomized controlled trial. A total of 60 patients scheduled for first-time CIED implantation will be randomized into two groups: the intervention group (SPSIPB with 30 mL 0.25% bupivacaine) and the control group (sham injection with 1 mL saline). All procedures will be performed under standard local anesthesia. The primary outcome is perioperative pain assessed by VAS intraoperatively and at 3, 6, 12, and 24 hours postoperatively. Secondary outcomes include postoperative sleep quality (SQ-NRS) and both patient and clinician satisfaction (5-point Likert scale). The trial will provide evidence regarding the potential of SPSIP block to improve perioperative analgesia and patient-centered outcomes in CIED implantation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Scheduled for first-time cardiac implantable electronic device (CIED) implantation (pacemaker or ICD)
* Able to provide written informed consent
* Normal coagulation profile
* No local infection at the planned block site

Exclusion Criteria:

* Severe heart failure (NYHA class IV)
* Morbid obesity (BMI >35 kg/m²)
* Known allergy to local anesthetics (e.g., bupivacaine)
* Coagulopathy or ongoing anticoagulant therapy contraindicating regional block
* Local infection at injection site
* Psychiatric or neurologic disorders interfering with pain/sleep assessment
* Revision or replacement CIED implantation (not first-time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity assessed by Visual Analog Scale (VAS) | Intraoperative and postoperative at 3, 6, 12, and 24 hours
  Pain levels will be assessed using a 0-10 Visual Analog Scale (VAS), where 0 = no pain and 10 = worst imaginable pain. Scores will be recorded intraoperatively and at 3h, 6h, 12h, and 24h postoperatively.

SECONDARY OUTCOMES:
Sleep quality assessed by Sleep Quality Numeric Rating Scale (SQ-NRS) | 24 hours after surgery
  Sleep quality will be measured using the SQ-NRS, scored from 0 = excellent sleep to 10 = worst possible sleep. A score ≥6 indicates poor sleep quality.
Patient satisfaction with procedure | 24 hours after surgery
  Patients will rate their satisfaction with the procedure on a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied).
Clinician satisfaction with procedure | 24 hours after surgery
  Clinicians performing the procedure will rate their satisfaction on a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Erkalp, MD, Study Director — Istanbul University-Cerrahpasa, Cardiology Institute
Locations (1):
- Gozde Altun, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093